CLINICAL TRIAL: NCT04433637
Title: Effect of Listed Music With Motivational Video And Nutrition on Non-Stress Test and Anxiety Level of Mother: Randomized Controlled Clinical Research
Brief Title: Effect of Listed Music With Motivational Video And Nutrition on Non-Stress Test and Anxiety Level of Mother
Acronym: NST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gülçin NACAR, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: gulcin nacar
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Related
Keywords: Non Stress Test; Motivational Video; Music; Nutrition; State Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition Group (Experimental): Pregnant women in the first experimental group were provided to consume cake and fruit juice 30 minutes before the NST procedure.
  Interventions: Dietary Supplement: Cake + fruit juice
- Video Group (Experimental): The video, which contains information about the developments and changes occurring in the mother and the fetus during pregnancy, was watched for 15-20 minutes during the NST procedure, accompanied by music that provided relaxation.
  Interventions: Other: Video group
- Control Group (No Intervention): No intervention was applied to the pregnant women in the control group.

INTERVENTIONS:
Dietary Supplement: Cake + fruit juice — Cake+fruit juice experiment group, pregnant were allowed to consume fruit juice and cake, and it was expected that half an hour would pass after feeding to get NST.
  Arms: Nutrition Group
Other: Video group — Music with motivational video experimental group, pregnant women were provided with fruit juice and cake, and it was expected that half an hour would pass after feeding to get NST. During this waiting period, the researchers were informed about the development and changes in the body and the fetus specific to the gestational week and NST. Later, NST was applied, and during the procedure, the pregnant women were watched with music that provides relaxation with the video regarding the fetal development appropriate for the gestational week and changes in the mother.
  Arms: Video Group

SUMMARY:
Objective: The research was conducted to determine the effect of music and nutrition played together with motivational video on non-stress test (NST) result and mother's anxiety level.

Method: The study was conducted as a randomized controlled clinical trial. The sample of the study consisted of 360 pregnant women, two experimental and one control group (120 pregnant women in each). In the study, pregnant women in the first experimental group were provided to consume cake and fruit juice 30 minutes before the NST procedure. The second experimental group was provided to eat fruit juice and cake before NST, and the video created with a similar content was given about the developments and changes occurring in the mother and fetus during pregnancy, and was watched for about 15-20 minutes during the NST procedure accompanied by music that provided relaxation. The data of the study were collected by using the Participant Presentation Form, NST evaluation form and State Anxiety Inventory.

DETAILED DESCRIPTION:
Non Stress Test (NST) has been used frequently in fetal health assessment in recent years due to its easy application, cheapness, reliability and rapid assessment. False negativity rates of NST also cause an increase in cesarean rates. Studies in recent years show that there are methods and factors that increase fetal movements and shorten NST application time. It was observed that nutrient intake, music playing, fetal acoustic vibration application and halogen light applications before NST increased fetal movements and shortened NST time.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or over
* Being pregnant more than 32 weeks gestation,
* Having at least one live birth,
* Having had NST before,

Exclusion Criteria:

* Having any risk factor (preeclampsia, IUGG, early membrane rupture, getational diabetes etc.) during pregnancy
* Urinary contraction after NST,
* It is a cardiovascular disease diagnosed in the fetus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 360 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Effect of nutrition | 1 month
  questionnaire NST Findings Registration Form
  As Reactive NST; The test result was accepted as reactive NST in the presence of at least two accelerations, which lasted at least 15 seconds within the 20-minute period when the electronic fetal heartbeat traces were printed and was 15 beats / minute more than the baseline beat.
  As nonreactive NST; The absence of at least two accelerations, which lasted at least 15 seconds within the 20-minute period when the electronic fetal heartbeat traces were printed, was 15 beats / minute more than the baseline beat, or 160 beats / minute and above continuous fetal tachycardia in the presence of severe variable decelerations and late decelerations. In case of development, the result was evaluated as nonreactive NST.
Effect of music with motivational video | 1 month
  scale State Anxiety Scale The state anxiety part of the scale consisting of two parts was used. Answer options on both scales consisting of twenty questions can get points from 1 to 4.
  There are direct and inverted expressions in the scales. Direct expressions express negative emotions, and reversed expressions express positive emotions. There are ten reversed expressions in the WHO and these are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The total score value obtained from the scale varies between 20 and 80. The increase in the score obtained from the scale indicates that the level of anxiety is high.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin N NACAR, PhD, Principal Investigator — İnönü Üniversitesi
Locations (1):
- Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taşhan ST, Çoşkun Eİ, Nacar G, Erci B. Effect of Listed Music With Motivational Video And Nutrition on Non-Stress Test and Anxiety Level of Mother: Randomized Controlled Clinical Research. Complementary Therapies in Medicine....